CLINICAL TRIAL: NCT05317338
Title: Effects of a Multicomponent Exercise Program on the Functional Performance and Cognitive Ability of Hospitalized Older People: A Randomized Clinical Trial
Brief Title: Multicomponent Exercises in Functional Performance and Cognitive Ability of Hospitalized Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-0119
Record Dates: First submitted 2021-12-08; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Old Age; Debility
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants randomized to this group will be enrolled to a multicomponent training for 5-7 consecutive days and will continue to receive usual hospital care. The training program consists of strength, balance and gait exercises performed within the hospital.
  Interventions: Behavioral: Group-based exercise training during hospitalization
- Control group (No Intervention): Participants randomized to the control group will receive only the usual hospital care and rehabilitation, without performing multicomponent exercises.

INTERVENTIONS:
Behavioral: Group-based exercise training during hospitalization — Multicomponent exercises for 5-7 days with acutely hospitalized older.
  Arms: Intervention group

SUMMARY:
Older patients spend most of their time in situations of muscle disuse during acute hospitalization. Physical inactivity is a key factor for the development of adverse events caused by hospitalization, known as iatrogenic nosocomial disability. Adopting a multicomponent training program during acute hospitalization can be an efficient strategy to reduce adverse effects and promote improvements in older health. This study is a randomized clinical trial with acutely hospitalized older individuals. Patients will be randomized into intervention and control groups. The intervention group will perform multicomponent training for 5-7 consecutive days, and will continue to receive usual hospital care. The control group will receive only the usual care and rehabilitation.

DETAILED DESCRIPTION:
This study is a randomized controlled trial with acutely hospitalized older individuals. The first aim is to evaluate the effects of a multicomponent training intervention on functionality, cognitive ability and inflammatory profile in older patients during acute hospitalization.

The population studied will be older patients (≥ 70 years), admitted to the Internal Medicine sector of the Hospital de Clinicas de Porto Alegre. The number of older people obtained through sample calculation is 30 individuals per group, totaling 60 participants in the study.

Patients will be randomized into intervention and control groups. The intervention group will perform multicomponent training for 5-7 consecutive days, and will continue to receive usual hospital care. Exercises aimed at the lower and upper limbs will be performed, such as sitting and standing up from a chair, leg press, bilateral knee extension and bench press with elastic tape. Balance and gait exercises will also be performed. The training session will be considered complete if patients are able to perform 90% or more of the scheduled exercises, the frequency and possible adverse events will be documented in daily records. The control group will not receive multicomponent physical training, only the usual care provided by the hospital. Both groups will be evaluated before and after 5-7 days of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 70 years and older;
* Able to tolerate exercise;
* Barthel Index ≥60;
* Be able to walk alone or with the aid of a cane, crutch or walkers;
* Be able to communicate and inform consent to participate in the research.

Exclusion Criteria:

* Length of stay <5 days;
* Inability to participate in the testing procedures and/or the multi-component training program, as determined by the physician;
* Present one or more factors:

  1. Terminal illness;
  2. Myocardial infarction in the last 3 months;
  3. Unstable cardiovascular disease;
  4. Any type of fracture in the last 3 months, which makes it impossible to carry out the movements;
  5. Severe dementia.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes in functional independence scores | Pre and post intervention (after 7 days), 1 and 3 months after hospital discharge.
  By using the Barthel Index. This tool indicates an individual's ability to perform basic activities of daily living. Scores range from 0 (severe functional dependence) to 100 (functional independence).
Changes in lower limbs functional capacity | Pre and post intervention (after 7 days), 1 and 3 months after hospital discharge.
  By using the Short Physical Performance Battery (SPPB) the mobility of the lower limbs will be evaluated through static balance tests while standing, walking speed and muscle strength

SECONDARY OUTCOMES:
Handgrip strength | Baseline and after the intervention period (after 7 days)
  Assessed using a handgrip dynamometer
Maximum dynamic muscle strength of lower limbs | Baseline and after the intervention period (after 7 days)
  Maximum strength assessed through the one repetition maximum test in the leg press and knee extension exercises.
Lower limb muscle power | Baseline and after the intervention period (after 7 days)
  Muscle power will be assessed in leg press and knee extension exercises, with intensities of 30% and 60% using an encoder device.
Walking ability | Baseline and after the intervention period (after 7 days)
  6 meter walking ability
Inflammatory markers | Baseline and after the intervention period (after 7 days)
  The following markers will be collected: C-reactive protein, leptin, tumor necrosis factor, interleukin, interferon, insulin like growth factor, transforming growth factor
Changes in cognitive state | Baseline and after the intervention period (after 7 days)
  The Mini Mental State Assessment instrument will be used. Questionnaire with a scale of 0 to 30 points, with 0 being the worst and 30 the best.
Changes in quality of life scores | Baseline and after the intervention period (after 7 days)
  Quality of life will be assessed using the EuroQol-5 Dimension questionnaire. Questionnaire that encompasses 5 health domains (mobility, personal care, usual activities, pain/discomfort and anxiety/depression) whose variation from 0 to 100 corresponds, respectively, to the worst and best health status.
Mortality | Pre and post intervention (after 7 days), 1 and 3 months after hospital discharge.
  Days alive since admission to hospital
Clinical condition | Pre and post intervention (after 7 days), 1, 3 and 12 months after hospital discharge.
  Information will be collected about clinical conditions (number of days of hospitalization and readmission).
Muscle thickness | Baseline and after the intervention period (after 7 days)
  The quadriceps muscle thickness will be evaluated by ultrasonography
Muscle quality | Baseline and after the intervention period (after 7 days)
  The muscle quality of the quadriceps will be evaluated through echo intensity using an ultrasound device
Changes in executive function | Baseline and after the intervention period (after 7 days)
  To assess executive function, the Trail Making Test will be performed
Level of agitation, sedation and delirium | Baseline and after the intervention period (after 7 days)
  The Confusion Assessment Method will be used
Changes in the depressive symptoms scale | Baseline and after the intervention period (after 7 days)
  The Geriatric Depression Symptoms (GDS) tool will be used. Score from 0 to 15, if greater than 5, the patient is suspected of having depression.

CONTACTS AND LOCATIONS:
Overall Officials: Emílio H Moriguchi, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No